CLINICAL TRIAL: NCT01948128
Title: A Phase 2 Randomized, Double-blind, Window of Opportunity Trial Evaluating Clinical and Correlative Effects of Vitamin D in Patients With Breast Cancer. The ICARUS Trial
Brief Title: Effects of Vitamin D in Patients With Breast Cancer
Acronym: OTT 12-06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120362-2OH
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Experimental): Vitamin D3 40,000 iu per day by mouth
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): Placebo taken daily by mouth
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Participants will take 4 capsules of Vitamin D which equals 40,000 IU by mouth daily during the wait time between diagnosis and surgery.
  Other Names: Vitamin D; cholecalciferol
  Arms: Vitamin D3
Other: Placebo — Participants will take 4 capsules of placebo by mouth daily during the wait time between diagnosis and surgery.
  Arms: Placebo

SUMMARY:
This protocol is a randomized, phase 2 "window of opportunity" trial assessing the biological effects of short term oral vitamin D administration on breast cancer clinical and translational markers in patients awaiting surgery at the Ottawa Hospital. It takes advantage of the current wait times (2-8 weeks) for breast cancer surgery as a "window of opportunity" to rapidly assess biological changes with vitamin D intake.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed female primary breast cancer patients whose surgery is planned for the next 2-8 weeks without neoadjuvant therapy as assessed by multidisciplinary team
2. Age ≥18 years
3. Clinically palpable tumour(s) (greater than or equal to 2 cm)
4. Normal serum and urine calcium and serum PTH values at baseline (as defined by Ottawa Hospital)
5. Written informed consent for study

Exclusion Criteria:

1. Patients with recurrent or metastatic breast cancer
2. History of neoadjuvant hormonal therapy, chemotherapy, or radiation therapy in the last 6 months for their breast cancer or any other cancer treatment
3. ECOG performance Status > 2
4. Hypercalciuria on initial baseline urine, defined as Ca/Creatinine Ratio> 1.0
5. Current or previous history of urolithiasis or hyperparathyroidism
6. Abnormal hepatic function according to Ottawa Hospital norms (Total Bilirubin >2x upper limit of normal, ALT/AST >3x upper limit of normal)and/or abnormal renal function (Creatinine > 150 µmol/L)
7. History of granulomatous disease such as tuberculosis or sarcoidosis.
8. Intake of Vitamin D (cholecalciferol) supplement ≥ 2000 IU/day within the last 2 months
9. Inability to comply with a study protocol in the opinion of the investigator (such as abuse of alcohol, drugs or psychotic states).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pre and post vitamin D administration Ki67 levels and Caspase 3 levels (as assessed according to the apoptosis assay) | baseline and 2-8 weeks from baseline
  Participants will have Ki67 and Caspase 3 levels performed on the tissue that was used to initially diagnose breast cancer. Those levels will then be compared to the tissue acquired at the time of surgery which will occur 2-8 weeks from diagnosis.

SECONDARY OUTCOMES:
Serum levels of 25-0HD and in vivo breast (cancer and non cancer) tissue levels of 1,25(OH) | Baseline and 2-8 weeks from baseline at the time of surgery
  Participant will have Serum levels of 25-0HD and in vivo breast cancer tissue levels of 1,25(OH) taken at baseline and surgery

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arnaout, Dr., Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Woman's Breast Health Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Arnaout A, Robertson S, Pond GR, Vieth R, Jeong A, Hilton J, Ramsey T, Clemons M. Randomized window of opportunity trial evaluating high-dose vitamin D in breast cancer patients. Breast Cancer Res Treat. 2019 Nov;178(2):347-356. doi: 10.1007/s10549-019-05392-9. Epub 2019 Aug 9. PMID 31399931